CLINICAL TRIAL: NCT02559037
Title: Effect of Acupuncture on Maintaining Active Crohn's Disease Intestinal Homeostasis Via Intestinal Microbiota and Peripheral Immunity: a Randomized Controlled Trial
Brief Title: Acupuncture Treatment for Active Crohn's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Institute of Acupuncture, Moxibustion and Meridian (Other)
Collaborators: Fudan University (Other); Shanghai University of Traditional Chinese Medicine (Other); Shanghai Jiao Tong University School of Medicine (Other); Indiana University School of Medicine (Other); Changhai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZYS2015-02
Record Dates: First submitted 2015-04-16; First posted 2015-09-24 (Estimated); Last update posted 2020-04-07 (Actual); Status verified 2019-12

CONDITIONS: Crohn's Disease
Keywords: acupuncture; moxibustion; intestinal microbiota; Peripheral immunity; Brain functional and structural changes
MeSH Terms: conditions — Crohn Disease | interventions — Acupuncture Therapy; Moxibustion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupuncture-moxibustion group (Experimental): Receiving acupuncture and moxibustion treatment.
  Interventions: Device: Acupuncture and moxibustion
- Sham acupuncture-moxibustion group (Sham Comparator): Receiving sham acupuncture and sham moxibustion.
  Interventions: Device: Sham acupuncture and moxibustion

INTERVENTIONS:
Device: Acupuncture and moxibustion — Acupuncture acupoints: CV12, bilateral ST36, ST37, SP6, SP9, SP4, LR3 and LI3. Disposable acupuncture auxiliary device and 0.30*40mm or 0.30*25mm acupuncture needles (hwato, suzhou medical supplies factory co., LTD.) were used. The needles were directly inserted 20-30mm into the skin and elicited a de-qi sensation. The needle was kept for 30 min.
  Moxibustion acupoints: bilateral ST25 and ST36. Using mild-warm moxibustion, The surface temperature of acupoints were maintained at 43 ℃ ± 1 ℃, 30min for each acupoint. Moxibustion and acupuncture were performed at the same time, once every other day, three times a week, a total of 12 weeks of treatment. After the treatment, subjects were followed up in the weeks 24, 36 and 48.
  Arms: Acupuncture-moxibustion group
Device: Sham acupuncture and moxibustion — The acupoints used are same to the experimental group. Same disposable acupuncture auxiliary device and 0.35 * 40mm acupuncture needle (flat and blunt needle tip, Hwato, Suzhou Medical Supplies Factory Co., Ltd.) was selected. When the needle was pricked to the acupoint, it did not penetrating into the skin. The subject only felt slight pain and do not have the de-qi sensation.
  Sham moxibustion : by using the same moxa stick, The surface temperature of acupoints were maintained at 37 ℃ ± 1 ℃, 30min for each acupoint. Sham acupuncture and sham moxibustion were performed at the same time. They were treated once every other day, three times a week, a total of 12 weeks. After the treatment, subjects were followed up in the weeks 24, 36 and 48.
  Arms: Sham acupuncture-moxibustion group

SUMMARY:
The purpose of this study is to observe the efficacy and safety of acupuncture and moxibustion for Crohn's disease and the regulation mechanism of intestinal microbiota and peripheral immunity.

DETAILED DESCRIPTION:
1. A randomized controlled trial.
2. Acupuncture and moxibustion treatment, placebo control.
3. To observe the efficacy and safety of acupuncture and moxibustion treatment versus placebo controlled for Crohn's disease.
4. To observe the effect on the regulation of intestinal microbiota in Crohn's disease.
5. To observe the effect on the regulation of peripheral immunity in Crohn's disease.
6. To observe the effect on the regulation of brain function and structure in Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

1. meet the diagnostic criteria of Crohn's disease;
2. age 16-70 years old;
3. patients with mild or moderate disease (150<CDAI<450) and evidence of active inflammation: serum C-reactive protein concentration ≥5 mg/L, fecal calprotectin concentration ≥250 μg/g, or obvious endoscopic evidence of ulcerations during the screening period of past 4 weeks;
4. patients who were not responsive, intolerant, dependent, or refused to use any one of the following medications: mesalazine, glucocorticoid, immunomodulator (azathioprine, methotrexate), and anti-TNF-α agents;
5. did not take or take one or more of the following drugs: prednisone <15 mg/d for at least one month, azathioprine (<1 mg/kg/d), methotrexate (<15 mg/week), or mesalazine (<4 g/d) for at least 3 months;
6. no history of use of anti-TNF-alpha or other biological agents within 3 months immediately preceding the enrolment in the study;
7. no previous history of receiving acupuncture;
8. provision of written informed consent.

Exclusion Criteria:

1. Pregnant or lactating women, and those desirous of conceiving in the near future;
2. patients with severe organic diseases;
3. patients with mental illness;
4. patients receiving antibiotics, probiotics, prebiotics, traditional Chinese medicine, or other drugs;
5. patients with multiple comorbid conditions that require long-term therapy with drugs, which may affect the outcome measures;
6. patients with severe extraintestinal manifestations, such as severe skin diseases, eye diseases, or thromboembolic diseases;
7. severe intestinal fistula, abdominal abscess, intestinal stenosis and intestinal obstruction, perianal abscess, gastrointestinal bleeding, bowel perforation, or other complications;
8. patients with short bowel syndrome;
9. patients with a history of abdominal or gastrointestinal surgery in the past six months;
10. patients with skin diseases or defects at the sites of acupuncture that prevents the application of acupuncture.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with clinical remission | Week 12
  Defined as Crohn's disease activity Index (CDAI) < 150 and decrease > 70

SECONDARY OUTCOMES:
The proportion of patients with clinical remission | Week 24, 36 and 48
  Defined as CDAI < 150 and decrease > 70
The proportion of patients with clinical response | Week 12, 24, 36 and 48
  Defined as CDAI decrease > 70
the mean change of CDAI from baseline | Week 12, 24, 36 and 48
  Difference in the mean change of CDAI from baseline between groups
Laboratory tests for disease activity | Week 12, 24, 36 and 48
  C-reaction protein, mg/L
Laboratory tests for disease activity | Week 12, 24, 36 and 48
  Erythrocyte sedimentation rate, mm/h
Laboratory tests for disease activity | Week 12, 24, 36 and 48
  blood platelet level, L
Quality of life on the Inflammatory Bowel Disease Questionnaire (IBDQ) | Week 12 and 24
  QOL assessment for Crohn's disease
Psychological factors on the Hospital anxiety and depression scale (HADS) | Week 12 and 24
  Anxiety and depression assessment for CD
The mean change of Crohn's disease endoscopic index of severity (CDEIS) | Week 48
  Intestinal inflammation performance
Fecal calprotectin tests for disease activity | Week 12
  Intestinal inflammation assessment
Histological scores for pathogenic manifestations | Week 48
  Hematoxylin-eosin staining and Histological scores
The proportion of clinical recurrences | Week 24，36 and 48
  Defined as CDAI > 150 and increased by ≥70 points or need to adjust drug to control active disease
Safety evaluation (Number of participants with treatment-related adverse events as assessed by CTCAE v4.0) | Week 12, 24，36 and 48
  Eg. acupuncture related bleeding, hematoma, fainting needle, etc; moxibustion related burns, blistering, etc
Subgroup analysis of the main outcome measure | Week 12
  Compare using chi square test with stratified method or Fisher's exact test, and Gender, BMI, CDAI score at baseline, concomitant medicine, Montreal classification, biologic use history, and surgical history were used as stratification factors.

OTHER OUTCOMES:
Intestinal microbiota | Week 12
  Fecal microbiota structure and diversity
Plasma inflammatory cytokine levels | Week 12
  IFN-γ, TNF-a, IL-1β IL-17,IL-23 etc.
Intestinal barrier function | Week 12
  Plasma Diamine oxidase，lipopolysaccharide, D-lactate level
Brain functional changes | Week 12
  Using fMRI (resting-state fMRI)
Brain structural changes | Week 12
  brain gray matter, white matter changes
Correlation analysis of the change of CRP level and intestinal flora and plasma inflammatory levels at the end of acupuncture treatment | Week 12
  To explore the relationship between CRP and intestinal flora and inflammation influenced by acupuncture
Correlation analysis of the change of CRP level and and brain structure and function | Week 12
  To explore the relationship between intestinal inflammation and brain function influenced by acupuncture
Correlation analysis of intestinal flora and brain structure and function | Week 12
  To explore the relationship between intestinal flora and brain-gut axis

CONTACTS AND LOCATIONS:
Overall Officials: Huangan Wu, MD,PhD, Study Chair — Shanghai University of TCM
Locations (1):
- Shanghai Institute of Acupuncture, Moxibustion and Meridian, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Bao C, Wu L, Wang D, Chen L, Jin X, Shi Y, Li G, Zhang J, Zeng X, Chen J, Liu H, Wu H. Acupuncture improves the symptoms, intestinal microbiota, and inflammation of patients with mild to moderate Crohn's disease: A randomized controlled trial. EClinicalMedicine. 2022 Feb 12;45:101300. doi: 10.1016/j.eclinm.2022.101300. eCollection 2022 Mar. PMID 35198926